CLINICAL TRIAL: NCT05406817
Title: A Phase 1, Open-label Study to Assess the Mass Balance, Pharmacokinetics, and Metabolism of Orally Administered [14C]-SNDX-5613 in Patients With Relapsed/Refractory Acute Leukemia
Brief Title: Study of Radiolabeled Revumenib in Adults With Acute Leukemia
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Syndax Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SNDX-5613-0705
Expanded Access: NCT05918913 (No longer available)
Record Dates: First submitted 2022-06-01; First posted 2022-06-07 (Actual); Last update posted 2025-01-10 (Actual); Status verified 2025-01

CONDITIONS: Acute Leukemia
Keywords: SNDX-5613; Acute Leukemia; Refractory leukemia; Relapsed leukemia
MeSH Terms: conditions — Leukemia | interventions — revumenib

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Revumenib (Experimental): Participants will be administered a single dose of revumenib (containing ~100 microcuries [14C]-revumenib) in the AME part of the study.
  Each dose administered after the first dose in the AME part of the study will be nonradiolabeled revumenib. revumenib may continue to be administered following completion of the AME part of the study. Doses will be administered in continuous 28-day cycles until either PD or unacceptable toxicity.
  Interventions: Drug: Revumenib

INTERVENTIONS:
Drug: Revumenib — Initial radiolabeled revumenib will be administered as an oral solution. Capsules will be administered thereafter.
  Other Names: SNDX-5613

SUMMARY:
This is an open-label study to evaluate the absorption, metabolism, and excretion (AME) of carbon-14 ([14C])-revumenib in participants with acute leukemia.

DETAILED DESCRIPTION:
Participants will be enrolled in this study primarily to complete the 11-day AME portion of the study; participants who are receiving benefit from revumenib may remain on study until progressive disease (PD) or unacceptable toxicity.

ELIGIBILITY:
Key Inclusion Criteria:

* Males and females (of non-childbearing potential) aged ≥18 years
* Relapsed or refractory acute leukemia, including participants who are MRD-positive by multiparametric flow cytometry or next-generation sequencing, and including participants with isolated extramedullary disease.
* Previously received standard of care therapy
* Eastern Cooperative Oncology Group (ECOG) performance status score of 0 to 2
* Adequate liver and cardiac function
* Fertile males agree to use barrier contraception from the time of enrollment through 120 days after the last study drug dose

Key Exclusion Criteria:

* Active diagnosis of acute promyelocytic leukemia
* White blood cell (WBC) count >25,000/microliters at time of enrollment.
* Detectable human immunodeficiency virus viral load within the previous 6 months
* Hepatitis B or Hepatitis C
* Cardiac, gastrointestinal, or graft-versus-host disease (GVHD)
* History of or any concurrent condition, therapy, laboratory abnormality, or allergy to excipients that might confound the results of the study, interfere with the participant's ability to participate for the full duration of the study, or not be in the best interest of the participant to participate
* Must not be receiving any moderate or strong cytochrome P450 3A4 (CYP3A4) inhibitor/inducers
* Any commercially available or investigational antileukemic therapy other than revumenib except for short-term administration of corticosteroids and/or hydroxyurea for cytoreduction
* Participation in another therapeutic interventional clinical study in which an investigational agent was administered within 30 days before starting revumenib
* Any concurrent systemic treatment to prevent GVHD

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2022-08-05 (Actual); Primary Completion 2024-11-18 (Actual); Study Completion 2024-11-18 (Actual)

PRIMARY OUTCOMES:
Percentage of Dose Excreted in Urine (feu) | Up to Day 11
Percentage of Dose Excreted in Feces (fef) | Up to Day 11
Amount Excreted in Urine (Aeu) | Up to Day 11
Amount Excreted in Feces (Aef) | Up to Day 11
Area Under The Concentration Time Curve from Time 0 to The Last Measurable Concentration (AUC0-t) | Up to Day 21
Maximum Observed Concentration (Cmax) | Up to Day 21

SECONDARY OUTCOMES:
Number of Participants with Treatment-emergent Adverse Events (TEAEs) | up to approximately 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Nicole McNeer, MD, PhD, Study Director — Syndax Pharmaceuticals
Locations (1):
- MD Anderson Cancer Center, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No